CLINICAL TRIAL: NCT04738656
Title: Mediterranean-style and Open Protein Diet Plans on Weight Loss in Patients With Obesity After Endoscopic Bariatric Treatment
Brief Title: Effectiveness of the Mediterranean Diet on Weight Loss After Endoscopic Bariatric Treatmen
Status: Completed | Type: Observational
Sponsor: Universitat Politècnica de Catalunya (Other)
Collaborators: University of Barcelona (Other); Clinica Dorsia (Unknown)
Responsible Party: Principal Investigator, Antonio Sanchez Egea, Assistant Professor, Universitat Politècnica de Catalunya
Other Study IDs: UPCatalunya
Record Dates: First submitted 2021-01-25; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Obesity; Obesity, Morbid
Keywords: Endoscopic bariatric treatment; Excess weight loss; Excess body mass index; Mediterranean diet plan; Open protein diet plan
MeSH Terms: conditions — Obesity; Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mediterranean-style diet plan: Mediterranean-style diet plan (6 months): 22% proteins, 53% carbohydrates, and 25% of lipids.
  52 participants.
  Interventions: Dietary Supplement: Diet plan
- Open protein diet plan: Open protein presents (6 months) 40% of proteins, 29% carbohydrate and 31% of lipids.
  26 participants.
  Interventions: Dietary Supplement: Diet plan

INTERVENTIONS:
Dietary Supplement: Diet plan — Mediterranean style is a non-restricted diet plan compared with the open protein diet plan

SUMMARY:
All participants were weighed every week for 24 weeks, wearing light clothes to the nearest 0.1 kg, using a body composition analyzer. Height was determined during the first clinic evaluation using a fixed wall stadiometer to the nearest 0.1 cm, in standing position.

Intervention: Participants followed a liquid diet plan during the first week after the endoscopic bariatric procedure (Bioenterics Intragastric Balloon - BIB - or Primary Obesity Surgery Endoluminal - POSE -). Subsequently, subjects were randomly assigned either a Mediterranean-style or a protein diet plan. Energy intake was calculated according to the Spanish Consensus on Bariatric Endoscopy.

The hypothesis of this project is to analyze whether the Mediterranean-style diet is more effective compared with the open protein diet plans in weight loss and weight relapse in subjects with obesity who underwent endoscopic bariatric therapies.

ELIGIBILITY:
Inclusion Criteria:

* no previous gastric intervention
* no hiatus hernias
* not being pregnant or in breastfeeding
* not having cardiac problems, and having regular values in coagulation and blood count,
* having a positive psychological evaluation.

Exclusion Criteria:

* lack of compliance with the dietary treatment
* adverse effects of the surgery
* refuse to complete the treatment
* lack of adherence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic. Patients of Dorsia Clinics Surgery and Aesthetic Medicine
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Weekly weight loss | Every week up to 24 weeks
Weight relapse after 36 weeks | 1 time after 36 weeks

IPD SHARING:
Plan to Share IPD: Undecided
By email: antonio.egea@upc.edu

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-01-25): https://cdn.clinicaltrials.gov/large-docs/56/NCT04738656/Prot_SAP_ICF_000.pdf